CLINICAL TRIAL: NCT06455124
Title: Short-course Radiotherapy Combined With CapeOx and PD-1 Inhibitor After Local Excision for High-risk Early Rectal Cancer (TORCH-LE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-31-3584
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Rectal Cancer
Keywords: early rectal cancer; high risk; local excision; radiation; PD-1 inhibitor; chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation; spartalizumab; toripalimab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): Patients will receive short course radiotherapy and four cycles of CapeOx and PD-1 inhibitor.
  Interventions: Radiation: Radiation; Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Radiation — Shor-course radiotherapy: 25Gy/5Fx
Drug: PD-1 antibody — PD-1 antibody (Toripalimab): 240mg d1 q3w
  Other Names: Toripalimab
Drug: Capecitabine — Capecitabine: 1000mg/m2 d1-14 q3w
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w

SUMMARY:
This is a single arm phase II study to explore the 3y LRFS and safety for high-risk early rectal cancer after local excision with short-course radiotherapy and chemo-immunotherapy.

DETAILED DESCRIPTION:
A total of 60 patients with high-risk pathologic stage pT1 or pT2 cancer after local excision but refused radical surgery will be included.

Eligibility criteria include a histological diagnosis of adenocarcinoma located ≤7 cm from the anal verge, pT1 after local excision of the primary rectal cancer, with one of the high-risk features including margin positivity/very close margin (<1mm) at time of local excision, depth of invasion >1 mm or SM3 invasion (submucosal invasion to the lower third of the submucosal level), high grade or poorly differentiated, lymphovascular invasion, perineural invasion, tumour budding, or pT2 tumor.

They will receive 5*5Gy short-course radiotherapy, followed by 4 cycles of capecitabine plus oxaliplatin (CAPOX) chemotherapy and PD-1 antibody.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years old, female and male
2. pathological confirmed adenocarcinoma
3. the distance from anal verge ≤ 7 cm
4. pT1 after local excision of the primary rectal cancer, with at least one of the high-risk features including margin positivity/very close margin (<1mm) at time of local excision, depth of invasion >1 mm or SM3 invasion (submucosal invasion to the lower third of the submucosal level), high grade or poorly differentiated, lymphovascular invasion, perineural invasion, tumour budding, or pT2 tumor.
5. refuse radical surgery
6. without pelvic or distance metastases
7. KPS >=70
8. with good compliance
9. microsatellite repair status is MSS/pMMR
10. without previous anti-cancer therapy or immunotherapy
11. signed the inform consent

Exclusion Criteria:

1. pregnancy or breast-feeding women
2. pathological confirmed signet ring cell carcinoma
3. history of other malignancies within 5 years
4. serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
5. immunodeficiency disease or long-term using of immunosuppressive agents
6. baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
7. DPD deficiency
8. allergic to any component of the therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
3y LRFS | From date of initiation of treatment until the date of first documented pelvic failure, assessed up to 36 months.
  Rate of 3 year local recurrence free survival rate

SECONDARY OUTCOMES:
3y DFS | From date of initiation of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Rate of 3 year disease free survival
3y OS | From date of initiation of treatment until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
Grade 3-4 adverse effects rate | From date of initiation of treatment until the date of death from any cause, assessed up to 36 months.
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the related article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 5 years following related article publication.
Access Criteria: Proposals should be directed to xxx@yyy. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link will to be included).